CLINICAL TRIAL: NCT01635465
Title: A Randomised Controlled Phase II Trial of Vinorelbine Plus Capecitabine Versus Docetaxel Plus Capecitabine in Anthracycline-pretreated Women With Metastatic Breast Cancer.
Brief Title: Vinorelbine Plus Capecitabine Versus Docetaxel Plus Capecitabine in Anthracycline-pretreated Women With Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIH-LSF-201205001
Record Dates: First submitted 2012-06-17; First posted 2012-07-09 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-07

CONDITIONS: Anthracycline-pretreated Metastatic Breast Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Observation group:vinorelbine plus capecitabine
- Control group:docetaxel plus capecitabine

SUMMARY:
Docetaxel plus Capecitabine in anthracycline-pretreated metastatic breast cancer is a recommended scheme in National Comprehensive Cancer Network (NCCN) guideline. Vinorelbine plus Capecitabine is also effective in Metastatic Breast Cancer (MBC) in some clinical study with small sample.

DETAILED DESCRIPTION:
A randomised controlled trial of vinorelbine plus capecitabine versus docetaxel plus capecitabine in anthracycline-pretreated women with metastatic breast cancer. The primary endpoints of the study is progression free survival (PFS). The secondary endpoints are overall response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* female ≥ 18 years old ECOG 0-2

Exclusion Criteria:

* brain metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 | -7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Li S, Meng W, Zhang J, Xie X, Hao C, Jia Y, Tong Z. A randomized controlled Phase II trial of vinorelbine plus capecitabine versus docetaxel plus capecitabine in anthracycline-pretreated women with metastatic breast cancer. J Cancer Res Ther. 2020 Sep;16(5):1069-1076. doi: 10.4103/jcrt.JCRT_792_19. PMID 33004749